CLINICAL TRIAL: NCT04407949
Title: Untersuchung Der Übereinstimmung Der Ereigniserkennung Von "prismaLine" Geräten Mit Der Polysomnographie
Brief Title: Comparison of Sleep Disordered Breathing Events Detected by the CPAP Device "prismaLine" With Polysomnography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: Heinen und Löwenstein GmbH & Co. KG (Industry)
Responsible Party: Principal Investigator, Georg Nilius, PD DR med, medical director of pneumologic department, Institut für Pneumologie Hagen Ambrock eV
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EventLab
Record Dates: First submitted 2019-09-13; First posted 2020-05-29 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Sleep Apnea Syndromes
Keywords: CPAP; Apnea; Hypopnea; event detection
MeSH Terms: conditions — Sleep Apnea Syndromes; Apnea | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Every enrolled patient underwent a CPAP - Titration under PSG with predefined pressure steps. Afterwards breathing events are scored manually based on AASM Criteria by a trained study member. The events will be compared with the readout from the CPAP Device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- event detection (Other)
  Interventions: Other: CPAP Treatment

INTERVENTIONS:
Other: CPAP Treatment — Comparing events from the CPAP device with the events scored in PSG
  Other Names: PrismaLine

SUMMARY:
Evaluation of residual sleep disordered breathing (SDB) under continuous positive airway pressure (CPAP) therapy with comparison of the automatic detected SDB event indices from CPAP machines with manual scored polysomnography (PSG).

DETAILED DESCRIPTION:
The evaluation of residual sleep disordered breathing (SDB) in sleep apnea (SA) after initiation of continuous positive airway pressure (CPAP) therapy is important to verify the therapeutic success. In clinical practice, the internal records of CPAP devices are utilized to determine the therapeutic success, during either medical consultations or telemetric observation.

This study was designed to evaluate the quality of SDB Event Indices (EI), which are recorded by the CPAP device (Prisma, Löwenstein Medical Technology).

The detected events of a manual scored polysomnography (PSG) in the sleep laboratory will be compared with the simultaneously recorded events of the CPAP device.

This shall lead to recommendations regarding the situations, and in which degree the event detection of the CPAP devices may be meaningful to determine the therapeutic success of home sleep apnea therapy.

ELIGIBILITY:
Inclusion Criteria:

* PSG diagnostic not older than 3 month,
* AHI>15, CPAP indication,
* age >18,
* nasal CPAP mask,
* written informed consent

Exclusion Criteria:

* CPAP contraindication,
* participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
apnea- hypopnea- index (AHI) | up to 8 hours
  Total number (N) and index (N/h) of sleep disordered breathing events (apnoeas plus hypopneas) from PSG and device log

SECONDARY OUTCOMES:
hypopnea index relating to oxygen desaturation | up to 8 hours
  total number of Hypopneas (N) and Index (N/h) scored under AASM criteria for hypopneas, both rules. 1A: hypopnea events with >= 3% oxygen desaturation and 1B: hypopnea events with >= 4% oxygen desaturation.
central and obstructive hypopnea index | up to 8 hours
  total number (N) and Index (N/h) of hypopneas scored under AASM criteria for central and obstructive hypopneas.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Kliniken Essen-Mitte, Evang. Huyssens-Stiftung/Knappschaft gGmbH
Locations (1):
- Kliniken Essen-Mitte, Evang. Huyssens-Stiftung/Knappschaft gGmbH, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richter M, Schroeder M, Domanski U, Schwaibold M, Nilius G. Reliability of respiratory event detection with continuous positive airway pressure in moderate to severe obstructive sleep apnea - comparison of polysomnography with a device-based analysis. Sleep Breath. 2023 Aug;27(4):1639-1650. doi: 10.1007/s11325-022-02740-w. Epub 2022 Nov 17. PMID 36394692